CLINICAL TRIAL: NCT03723863
Title: The Evaluation of a Work Intervention to Facilitate Work Maintenance or Re-Entry to the Workforce for Breast Cancer Patients
Brief Title: Occupational Therapist-Led Work Intervention in Facilitating Work Maintenance or Re-entry to the Workforce in Patients With Stage I to III Breast Cancer Undergoing Chemotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study team determined that data collected was appropriate for study outcome goals.
Sponsor: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RG1718049; NCI-2018-02059 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9993 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-10-23; First posted 2018-10-30 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Breast Cancer Stage I; Breast Cancer Stage III; Breast Cancer Stage II; Breast Cancer Stage IIA; Breast Cancer Stage IIB; Breast Cancer Stage IIIA; Breast Cancer Stage IIIB; Breast Cancer Stage IIIc; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Occupational Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (Occupational therapy) (Experimental): Patients receive in-person occupational therapist-led work consultation
  Interventions: Behavioral: Occupational Therapy

INTERVENTIONS:
Behavioral: Occupational Therapy — Receive in-person occupational therapist-led work consultation
  Other Names: Occupational Therapy, OT

SUMMARY:
This trial studies how well occupational therapy (occupational therapist-led work intervention) works in facilitating work maintenance or re-entry to the workforce for stages I to III breast cancer patients who will be undergoing curative intent chemotherapy. Occupational therapy may help cancer patients maintain employment or successfully return to work soon after treatment.

DETAILED DESCRIPTION:
Patients receive in-person occupational therapist-led work consultation.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III breast cancer patients who will be undergoing curative intent chemotherapy
* Working in a paid capacity (part or full-time) at time of diagnosis with the intent to maintain or return to work following treatment

Exclusion Criteria:

* Non-English speaking patients. This study requires completing online questionnaires that are written in English and will not be translated
* Patients with a psychiatric or neurological condition that impairs capacity to make decisions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Change in perceived work ability | Baseline up to 3 years
  Will be measured by the Work Abilities Index (WAI).

SECONDARY OUTCOMES:
Change in health related quality of life | Baseline up to 3 years
  Will be measured by the Functional Assessment of Cancer Therapy General (FACT-G), a validated measure for quality of life in patients with cancer.
Change in financial toxicity | Baseline up to 3 years
  Will be measured by the Comprehensive Score for Financial Toxicity (COST-FACIT), a validated measure for financial toxicity for clinically relevant patient-centered outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Yung, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No